CLINICAL TRIAL: NCT02078791
Title: Perception of Discomfort and Psychosocial Difficulties in People With Diagnosis of Fibromyalgia and Predominant Neck Pain
Brief Title: Discomfort and Psychosocial Difficulties in Fibromyalgia
Acronym: Fibroebre
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Collaborators: Catalan Institute of Health (Other Government); Universidad Nacional de Educación a Distancia (Other)
Responsible Party: Principal Investigator, Pilar Montesó Curto, Dr., University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012LINE-01
Record Dates: First submitted 2014-02-27; First posted 2014-03-05 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Group Problem Solving Technique; infiltration
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Botox infiltration (Experimental): Botox infiltration in cervical region
  Interventions: Drug: Botox infiltration
- Psychology therapy (Experimental): Problem solving group therapy
  Interventions: Behavioral: Psychology therapy
- Botox infiltration & psychology therapy (Experimental): Botox infiltration in cervical region and problem solving group therapy.
  Interventions: Other: Botox infiltration & psychology therapy

INTERVENTIONS:
Drug: Botox infiltration — botox cervical infiltration in a group
  Other Names: botox infiltration, and grup solving terapy group
  Arms: Botox infiltration
Behavioral: Psychology therapy — Psychology problem solving therapy lead by specialized nurses.
  Other Names: Problem solving group therapy
  Arms: Psychology therapy
Other: Botox infiltration & psychology therapy — Botox infiltration in cervical region and psychology problem solving therapy lead by specialized nurses.
  Other Names: Botox infiltration and problem solving group therapy.
  Arms: Botox infiltration & psychology therapy

SUMMARY:
The patients who were not pain control, are referred to the Chronic Pain Unit so its complexity is greater. Made two different interventions in three groups of people with fibromyalgia. In the first group will proceed to infiltrate the painful area with medication, in the second GPST (Group Problem Solving Technique) and the third group both techniques. GPST will want to identify problems that people associate with fibromyalgia, as well as proposed solutions and it they have been carried out successfully or not. Will be essential to identifying and solving problems and using techniques to increase assertiveness, self-esteem and eliminating negative thoughts. Observing if after performing any of these techniques (infiltration, GPST or both) there is a better quality of life, reduce thoughts of suicide, pain and improves sleep quality. We also analyzed the satisfaction or not with therapies received and perceived usefulness.

DETAILED DESCRIPTION:
It is a clinical trial. STUDY SUBJECTS. By random sampling will distribute women diagnosed with fibromyalgia in three groups. 30 people are expected to include in each of the three groups. Group 1. Infiltration, GPST Group 2, Group 3 GPST+ Infiltration The sample size is approximately 30 so that alpha risk of 0.05, and a lower risk beta 0.2, 29 subjects needed to detect a difference equal to or greater than 0.25 units. It is assumed that the proportion in the control group is 0.8. has estimated a loss rate of 20% follow-up.

Fibromyalgia patients attending the chronic pain unit referred by family doctors and other specialists. These are patients who have painful symptoms that could not be controlled in the first level of health care or health centers.Not form part of the study all patients with fibromyalgia but only those who have discomfort in the cervical area preferably.To include in the study the patient acceptance of its participation is required by informed consent.Anesthesiologists assigned patients into three different groups according to the intervention takes place; infiltration, TRP (Problem Solving Therapy) or both interventions. When patients have met 8-10 start TRP group. Each group will be directed by a trained professional nursing. If we if we haven't enough sample will search in Fibromyalgia Associations.

The information of all variables are entered into a database (Excel) of which will be imported to a statistical program (SPSS) for analysis.

Qualitative variables were expressed as frequencies and percentages and quantitative mediated by central tendency and (mean and standard deviation) dispersion.The relationship between variables was analyzed by the χ2, comparison of means (t-student), analysis of variance (ANOVA) and Spearman, depending on the type of variable.Multivariate analysis will be performed to try to determine factors that may promote improved quality of life / patients.

It is considered that the difference between variables is significant when the significance level is less than or equal to 0.05 (p ≤ 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosing Fibromyalgia.
* Diagnosing Fibromyalgia + other causative pathology of chronic pain (chronic and / or chronic low back pain neck pain).
* Acceptance of study participation by informed consent

Exclusion Criteria:

* Severe disability that makes a first indication infiltration (disc herniation and / or lumbar spinal stenosis).
* cognitive Impairment
* Life expectancy less than 12 months

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-07; Primary Completion 2013-09 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in pain perception Visual Analogical Scale (VAS) | Baseline and 2 months

SECONDARY OUTCOMES:
Change in suicidal thoughts Plutchick Scale | Baseline and 2 months
change in quality of sleep SCOPA questionnaire | Baseline and 2 months
Change in health questionnaire EQ5D5L | Baseline and 2 months

OTHER OUTCOMES:
Change in satisfaction and perceived usefulness questionnaire | Baseline and 2 months

CONTACTS AND LOCATIONS:
Overall Officials: PILAR MONTESÓ, phD, Study Director — University Rovira i Virgili
Locations (1):
- Hospital Verge de la Cinta, Tortosa, Tarragona, Spain

REFERENCES:
- See also: Click here for more information about this study: Clinical Trial of Fibromyalgya in Southern Catalonia — http://www.fibromyalgia.org